CLINICAL TRIAL: NCT06415383
Title: Testing the Effects of High-dose Vitamin B6 Supplements on Pain Thresholds and Tolerance in Healthy Adults
Brief Title: The Effects of Vitamin B6 Supplementation on Pain Thresholds and Tolerance
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: INNOPURE (Unknown)
Responsible Party: Principal Investigator, David Field, Associate professor, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UREC24/13
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-05

CONDITIONS: Pain
Keywords: Vitamin B6; GABA; Excitation-Inhibition balance
MeSH Terms: conditions — Pain | interventions — Vitamin B 6

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin-B6 (Experimental): Participants will consume one high-dose Vitamin B6 100 mg tablet orally once daily for one month. Vitamin B6 will be provided as Pyridoxal-5'-Phosphate (PLP).
  Interventions: Drug: Vitamin B6 100 MG
- Placebo (Placebo Comparator): Participants will consume a Placebo tablet matching the appearance of the Vitamin B6 tablets in the Experimental arm orally once daily for one month.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin B6 100 MG — Vitamin B6 in for the form of pyridoxal phosphate (PLP)
  Arms: Vitamin-B6
Other: Placebo — Placebo tablet containing microcrystalline cellulose
  Arms: Placebo

SUMMARY:
This clinical trial aims to explore the effect of Vitamin B6 supplementation on pain thresholds and tolerance in healthy adults using thermal and electrical stimulation. Researchers will compare a placebo group to high-dose Vitamin-B6 to see if vitamin B6 increases pain thresholds and tolerance.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

* How does vitamin B6 affect pain thresholds and tolerance following a single 100mg dose?
* How does vitamin B6 affect pain thresholds following daily supplementation for up to a month?
* Does vitamin B6 supplementation affect measures related to the experience of pain, such as state anxiety, sleep, diet, and mood at different time points

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years
* Fluent speaker of English language

Exclusion Criteria:

* Under 18 years
* Presence or history of chronic pain
* Presence of neuropathic/nerve pain
* Raynaud's syndrome
* Using any vitamin supplementations that contain Vitamin B6 at more than the RDA, or combinations of B vitamins.
* On any medication that is GABA agonistic
* Any use of analgesic/anti-inflammatory medication up to 48 hours prior to any of the testing sessions.
* Any heart conditions
* Newly acquired tattoos on the pain stimulation site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Thermal sensory threshold | This will be done at baseline, 4-5 hours, 3-5 days, 11-13, and 28-35 days after the start of the intervention
  Sensory threshold will be measured using thermal stimulation (heat stimulation). The starting temperature of the applied probe will be adjusted to the individual's skin temperature and then slowly increased (0.5 deg C/s) until the participant feels a slight warm sensation. For safety, the temperature will never exceed 50 deg C. The procedure will be repeated three times. The average change in temperature (in degree Celsius) needed for participants to perceive a warm sensation will be used as outcome measure. Low values will therefore indicate a high sensitivity to warmth, whereas high values will indicate a low warmth sensitivity.
Thermal pain threshold | This will be done at baseline, 4-5 hours, 3-5 days, 11-13, and 28-35 days after the start of the intervention
  Pain threshold will be measured using thermal stimulation (heat stimulation). The starting temperature of the applied probe will be adjusted to the individual's skin temperature and then slowly increased (1 deg C/s) until the participant feels a slight pain/burning sensation. For safety, the temperature will never exceed 50 deg C. The procedure will be repeated three times. The average change in temperature (in degree Celsius) needed for participants to perceive a slight pain/burning sensation will be used as outcome measure. Low values will therefore indicate high pain sensitivity, whereas high values will indicate low pain sensitivity.
Electrical pain sensitivity | This will be done at baseline, 4-5 hours, 3-5 days, 11-13, and 28-35 days after the start of the intervention
  Pain sensitivity will be measured using electrical stimulation. Starting at an initial intensity of 0.3 mA, the intensity of each subsequently applied electrical stimulus will be increased in steps of 0.3 mA each, with a maximum intensity of 10 mA. The procedure will be continued until the participant perceives the applied shock as moderately painful (equivalent to a pain rating of 5 out of 10 or higher). The procedure will be repeated three times. The average intensity (in mA) needed for participants to perceive a moderate pain sensation will be used as outcome measure. Low values will therefore indicate a high sensitivity to electrical stimulation, whereas high values will indicate a low pain sensitivity in response to electrical stimulation.
Thermal pain tolerance | This will be done at baseline, 4-5 hours, 3-5 days, 11-13, and 28-35 days after the start of the intervention
  Pain tolerance will be measured using thermal stimulation (heat stimulation). The starting temperature of the applied probe will be adjusted to the individual's skin temperature and then slowly increased (1 deg C/s) until the participant feels that they can't tolerate the heat anymore. For safety, the temperature will never exceed 50 deg C. The procedure will be repeated three times. The average change in temperature (in degree Celsius) needed for participants to reach their pain tolerance will be used as outcome measure. Low values will therefore indicate low pain tolerance, whereas high values will indicate high pain tolerance.
Cold immersion pain tolerance | This will be done at baseline, 3-5 days, 11-13, and 28-35 days after the start of the intervention
  Pain tolerance will be measured by recording the number of seconds the participant is willing to keep their hand immersed in a 5 degree celsius cold bath, up to a maximum of 120 sec.
Pain wind-up | This will be done at baseline, 4-5 hours, 3-5 days, 11-13, and 28-35 days after the start of the intervention
  Pain sensitisation will be measured using a wind-up paradigm (temporal summation) with thermal stimulation (heat simulation).
  The thermal probe will start at 32 deg C and increase in temperature (100 deg C/s) to 49 deg C. After a duration of 800 ms, the temperature will return to baseline. Participants will be asked for a pain rating on a scale form 0 (not painful) to 10 (extremely painful). Subsequently, a series of 10 heat stimuli (identical to the once above, ISI 400 ms) will be applied. Participants will be asked to rate the most intense pain that they felt across the series, using the same 0-10 rating scale. The difference in pain ratings in response to the series and to the single stimulus will be used as the outcome measure. Higher (positive) ratings will indicate a stronger sensitisation to repeated painful stimuli. In contrast, negative values will indicate habituation to repeated painful stimuli.

SECONDARY OUTCOMES:
State anxiety | This will be done at baseline, 4-5 hours, 3-5 days, 11-13, and 28-35 days after the start of the intervention
  State anxiety will be measured using the State-Trait Anxiety Inventory (STAI), which produces a minimum score of 20 and a maximum score of 80, where higher scores indicate greater anxiety.
Positive and negative affect | This will be done at baseline, 4-5 hours, 3-5 days, 11-13, and 28-35 days after the start of the intervention
  State positive and negative affect will be measured using the The Positive And Negative Affect Schedule Now (PANAS-N) (PANAS-N; adapted from Watson et al., 1988).
Sleep quality | This will be done at baseline, 3-5 days, 11-13, and 28-35 days after the start of the intervention
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI), which results in a score ranging between 0 and 21, where higher scores indicate worse sleep quality.
Dietary intake | This will be measured at baseline during their first visit only
  Dietary intake will be measured using the Mediterranean Diet Adherence Screener(MEDAS), which produces a score ranging between 0 and 14, where higher scores indicate greater adherence to the Mediterranean diet.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spielberger, C. D., Gonzalez-Reigosa, F., Martinez-Urrutia, A., Natalicio, L. F., & Natalicio, D. S. (1971). The state-trait anxiety inventory. Revista Interamericana de Psicologia/Interamerican journal of psychology, 5(3 & 4).
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Martinez-Gonzalez MA, Garcia-Arellano A, Toledo E, Salas-Salvado J, Buil-Cosiales P, Corella D, Covas MI, Schroder H, Aros F, Gomez-Gracia E, Fiol M, Ruiz-Gutierrez V, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Munoz MA, Warnberg J, Ros E, Estruch R; PREDIMED Study Investigators. A 14-item Mediterranean diet assessment tool and obesity indexes among high-risk subjects: the PREDIMED trial. PLoS One. 2012;7(8):e43134. doi: 10.1371/journal.pone.0043134. Epub 2012 Aug 14. PMID 22905215